CLINICAL TRIAL: NCT05197283
Title: Determining the Effect of Three Types of Spaghetti (Regular, Whole Wheat and High Fiber-low Carbohydrates) on Glycemic Responses in Healthy Humans
Brief Title: Determining the Glycemic Effects of Three Types of Spaghetti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HRBD 49 11/10/2021
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
Keywords: blood glucose; spaghetti; glycemic index; glycemic load
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Investigator
Masking Description: single blind (investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Glucose as reference food (Experimental): Fourteen healthy, normal body weight adults (male: 6, female: 10) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested two times, in different visits as reference food; and 50g available carbohydrates from white bread, tested two times; and 50 gr available carbohydrates from spaghetti No7 types, regular, whole wheat and low carbohydrates - high fibre, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose and salivary insulin sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Other: Regular spaghetti; Other: Whole wheat spaghetti; Other: High fibre - low carbohydrates spaghetti
- White bread (Experimental): Fourteen healthy, normal body weight adults (male: 6, female: 10) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested two times, in different visits as reference food; and 50g available carbohydrates from white bread, tested two times; and 50 gr available carbohydrates from spaghetti No7 types, regular, whole wheat and low carbohydrates - high fibre, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose and salivary insulin sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Other: Regular spaghetti; Other: Whole wheat spaghetti; Other: High fibre - low carbohydrates spaghetti
- Regular spaghetti No 7 (Experimental): Fourteen healthy, normal body weight adults (male: 6, female: 10) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested two times, in different visits as reference food; and 50g available carbohydrates from white bread, tested two times; and 50 gr available carbohydrates from spaghetti No7 types, regular, whole wheat and low carbohydrates - high fibre, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose and salivary insulin sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Other: Regular spaghetti; Other: Whole wheat spaghetti; Other: High fibre - low carbohydrates spaghetti
- Whole wheat spaghetti (Experimental): Fourteen healthy, normal body weight adults (male: 6, female: 10) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested two times, in different visits as reference food; and 50g available carbohydrates from white bread, tested two times; and 50 gr available carbohydrates from spaghetti No7 types, regular, whole wheat and low carbohydrates - high fibre, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose and salivary insulin sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Other: Regular spaghetti; Other: Whole wheat spaghetti; Other: High fibre - low carbohydrates spaghetti
- High fiber - low carbohydrate spaghetti (Experimental): Fourteen healthy, normal body weight adults (male: 6, female: 10) after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested two times, in different visits as reference food; and 50g available carbohydrates from white bread, tested two times; and 50 gr available carbohydrates from spaghetti No7 types, regular, whole wheat and low carbohydrates - high fibre, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose and salivary insulin sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Other: Regular spaghetti; Other: Whole wheat spaghetti; Other: High fibre - low carbohydrates spaghetti

INTERVENTIONS:
Other: Glucose as reference food — Fourteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g glucose diluted in 300ml water, tested two times, in different visits, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: White bread — Fourteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from white bread, along with 300ml water, tested two times, in different visits, within 10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Regular spaghetti — Fourteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from regular spaghetti No 7, along with 300ml water, tested once, within 10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Whole wheat spaghetti — Fourteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from whole wheat spaghetti No 7, along with 300ml water, tested once, within 10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: High fibre - low carbohydrates spaghetti — Fourteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from high fibre - low carbohydrate spaghetti No 7, along with 300ml water, tested once, within 10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.

SUMMARY:
This study investigated the effects of thee types of spaghetti No7 on the glycemic response

DETAILED DESCRIPTION:
This study aimed to 1. determine the glycemic index and glycemic load of thee spaghetti No7 types (regular, whole wheat and high fiber-low carbohydrates) and 2. investigate the effects of these spaghetti types on postprandial glycemic response in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* non-diabetic men and women
* body mass index between 18 and 25 kg/m2

Exclusion Criteria:

* severe chronic disease (e.g. cardiovascular diseases, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* gastrointestinal disorders
* pregnancy
* lactation
* competitive sports
* alcohol abuse
* drug dependency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test

SECONDARY OUTCOMES:
Salivary insulin responses | 2 hours
  Clinically useful change in salivary insulin, defined as the restoration of insulin within normal limits during the 2hr glucose tolerance test
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in the form of booklet, one scale per page) at baseline, 15, 30, 45, 60, 90 and 120min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g. hunger, satiety, desire to eat etc
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure before and 2hr after consumption of the spaghetti products

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No